CLINICAL TRIAL: NCT03909308
Title: Effects of a Beach Tennis Training Session on Ambulatory Blood Pressure in Hypertensive Individuals: a Randomized Clinical Trial
Brief Title: Beach Tennis And Hypertension Study
Acronym: BAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 96487118000005327a
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
Keywords: Exercise; Beach Tennis; Sport training; Post exercise hypotension; Ambulatory blood pressure monitoring
MeSH Terms: conditions — Hypertension; Motor Activity; Post-Exercise Hypotension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control session (No Intervention): Control session without any exercise. The participants remained in seated rest throughout 45 min.
- Beach Tennis session (Experimental): The participants performed a beach tennis training session throughout 45 min.The session started with a standardized 5-minute warm-up consisting of basic techniques (i.e., serve, volley, forehand, and backhand) followed by three 12-minute beach tennis matches with 2-minute intervals between the games. We used regular beach tennis rules in the game, which was played on a regular beach tennis court (i.e., 16 m long by 8 m wide and net 1.70 m high).
  Interventions: Behavioral: Beach Tennis session

INTERVENTIONS:
Behavioral: Beach Tennis session — The Beach Tennis training session will be composed by a warm up of 5 min of BT in which technical exercises (i.e., serve, volley, forehand and backhand) will be performed After that, 3 BT small games of 12 min with a 2 minute interval between games using the conventional rules of sport will be performed. Before the session and after each small game, data regarding heart rate, blood pressure and rate perceived exertion will be recorded.
  Arms: Beach Tennis session

SUMMARY:
The purpose of the present study was to evaluate the effect of a beach tennis session on 24-hour ambulatory blood pressure in adults with hypertension. The main hypothesis is that a single session of beach tennis would decrease ambulatory blood pressure compared with a non-exercise control session.

DETAILED DESCRIPTION:
In this randomized crossover trial, participants performed randomly assigned two experimental sessions: a beach tennis session and a non-exercise control session. The beach tennis session started with a standardized 5-minute warm-up consisting of basic techniques, followed by three 12-minute beach tennis matches with 2-minute intervals between them. Heart rate and rating of perceived exertion were continuously recorded during the beach tennis session, and enjoyment was measured after the beach tennis session. The control session was performed in seated rest. Both experimental sessions lasted 45 minutes. Ambulatory blood pressure was measured continuously for 24-hour after sessions.

ELIGIBILITY:
Inclusion Criteria:

* Office blood pressure between 130-179 and 80-110 mmHg for systolic and diastolic blood pressure, respectively;
* Non-engaged in structured exercise programs in the last 3 months before the beginning of this study;
* Able to perform the proposed exercises.

Exclusion Criteria:

* Underlying cardiovascular disease in the last 24 months such as acute myocardial infarction, angina, stroke or heart failure;
* Diseases that reduce life expectancy;
* Smokers;
* BMI >39.9 kg/m²;
* Diabetic proliferative retinopathy.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Ambulatory Blood Pressure | 24 hours after control and beach tennis sessions
  Day-time, night-time and 24h ambulatory blood pressure measured through automatic oscillometric device after 45 min of control session and beach tennis session

SECONDARY OUTCOMES:
Systolic blood pressure | 45 minutes
  Systolic blood pressure in mmHg will be measured using automatic oscillometric before and after each experimental session throughout 45 min.
Diastolic blood pressure | 45 minutes
  Diastolic blood pressure in mmHg will be measured using automatic oscillometric before and after each experimental session throughout 45 min.
Blood Pressure Variability | 24 hours
  Systolic and diastolic BP values obtained in the 24-hour ambulatory blood pressure monitoring, with valid measures included in a programmed software to calculate the average real variability of these measures.
Enjoyment (PACES questionnaire) | 5 minutes
  Enjoyment will be measured after beach tennis session, the scale is composed of 18 items in a bipolar affirmations format (i.e., "amused" versus "not-amused") punctuated in a range from the minimum value "1" to the maximum value "7".

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ferrari, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Domingues LB, Carpes LO, Fuchs SC, Ferrari R. Effects of a single beach tennis session on short-term blood pressure variability in individuals with hypertension: a randomized crossover trial. Blood Press Monit. 2022 Jun 1;27(3):185-191. doi: 10.1097/MBP.0000000000000586. Epub 2022 Mar 7. PMID 35258025
- [Derived] Carpes L, Jacobsen A, Domingues L, Jung N, Ferrari R. Recreational beach tennis reduces 24-h blood pressure in adults with hypertension: a randomized crossover trial. Eur J Appl Physiol. 2021 May;121(5):1327-1336. doi: 10.1007/s00421-021-04617-4. Epub 2021 Feb 15. PMID 33590342